CLINICAL TRIAL: NCT05429008
Title: A Phase I, Multicenter, Open-label Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of HMPL-A83 in Patients With Advanced Malignant Neoplasm
Brief Title: A Phase I Clinical Study of HMPL-A83 in Patients With Advanced Malignant Neoplasm
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-A83-00CH1
Record Dates: First submitted 2022-06-14; First posted 2022-06-23 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Advanced Tumors
Keywords: CD47, HMPL-A83

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HMPL-A83 (Other): Drug: HMPL-A83 The starting dose of HMPL-A83 is 0.3 mg/kg IV QW with escalating dose levels of 1, 3, 10, 20, and 30 mg/kg IV QW, in 28-day treatment cycles.
  During the study, the below dose had also been selected: 10,20, and 30 mg/kg Q2W in 28-day treatment cycles; 30 and 45mg/kg Q3W.
  Interventions: Drug: HMPL-A83 injection

INTERVENTIONS:
Drug: HMPL-A83 injection — Day 1,8,15,22 dose; 28 day treatment cycles.
  Other Names: HMPL-A83

SUMMARY:
This is an open-label, first-in-human (FIH) Phase I study to evaluate the safety, tolerability, and preliminary efficacy of a humanized anti-CD47 monoclonal antibody (HMPL-A83) in patients with advanced malignant neoplasm.

DETAILED DESCRIPTION:
This is an open-label, first-in-human (FIH) Phase I study to evaluate the safety, tolerability, and preliminary efficacy of a humanized anti-CD47 monoclonal antibody (HMPL-A83) in patients with advanced malignant neoplasm. The sample size of this study is mainly based on the design of classical 3 + 3 combined accelerated titration dose escalation with a total of 6 dose groups, and approximately 31-84 patients are expected to be enrolled. During the dose escalation, DLT-nonevaluable patients will be replaced, or the actual number of patients enrolled may exceed the planned one due to adjustment of escalation schedule during the dose escalation. It is expected that no more than 99 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Solid tumors/lymphomas/AML/MDS with confirmed per study protocol;
2. Is willing and able to provide informed consent;
3. Aged 18-75 years (inclusive);
4. Life expectancy ≥12 weeks as judged by the investigator;
5. Female patients of childbearing potential and male patients with partners of childbearing potential agree to use a highly effective form(s) of contraception per study protocol.

Exclusion Criteria:

1. Previous exposure to any agent targeting the CD47/SIRP alpha axis.
2. Those concurrently participating in another interventional clinical study, excluding those concurrently participating in an observational (non-interventional) clinical study, or in the survival follow-up phase of an interventional study.
3. Those have received any investigational drug within 4 weeks prior to the first dose of study drug (note: investigational drug refers to the drug that has not been approved for marketing in China).
4. Those with prior anti-tumor therapy-induced toxicity (excluding alopecia or fatigue) not recovered to Grade 0 or 1 as defined by NCI CTCAE v5.0, including immune-related adverse events (irAEs) that have not recovered following immunotherapy, prior to the first dose of study treatment (≥ 4 weeks);
5. Those expected to require other systemic anti-tumor therapies such as chemotherapy, immunotherapy, biotherapy, or hormonal therapy (except palliative radiotherapy) during the study.
6. Those who have received prior immunotherapy such as anti-PD- (L) 1 antibody and discontinued due to ≥ Grade 3 irAEs.
7. Those with known hereditary or acquired bleeding disorder; uncontrolled active bleeding, coagulopathy; prior history of chronic haemolytic anaemia or positive hemolysis test at screening.
8. Patients with a history of deep venous thrombosis, pulmonary embolism, or any other serious thromboembolism within two years prior to enrollment, or those currently requiring anticoagulant or thrombolytic therapy as a therapeutic use.
9. Those have received immunosuppressive drugs within 4 weeks prior to the first dose of study drug
10. Those requiring long-term systemic hormonal therapy or any other immunosuppressive medication (excluding inhaled corticosteroid therapy or treatment at equivalent physiological doses).
11. Those have received live attenuated vaccines within 4 weeks prior to the first dose of study drug or planned to receive live attenuated vaccines during the study (for solid tumors)/any type of vaccine (for lymphoma, AML, MDS).
12. Those who have received any major surgical operation or uncured wound, ulcer or bone fracture within 4 weeks prior to the first dose of study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
safety information/AE,SAE | up to 3 years
  To evaluate the safety and tolerability of HMPL-A83 in patients with advanced tumors
MTD and RP2D | up to 2 years
  To determine the maximum tolerated dose (MTD) and/or the recommended phase II dose (RP2D) of HMPL-A83 in patients with advanced tumors.

SECONDARY OUTCOMES:
PK endpoints | up to 3 years
  To investigate the pharmacokinetic (PK) profile of HMPL-A83 in patients with advanced tumors, including but not limited to the maximum plasma concentration (Cmax), trough concentration (Ctrough or Cmin), elimination half-life (t1/2), area under the plasma concentration-time curve (AUC0-t, AUC0-∞, AUC0-τ), apparent clearance (CL), apparent volume of distribution at steady state (Vss), etc.
Efficacy endpoints | up to 3 years
  objective response rate (ORR)

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, Principal Investigator — Shanghai East Hospital
Locations (4):
- China (4):
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shandong Cancer Hospital, Shandong, Jinan
  - Shanghai Orient Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No